CLINICAL TRIAL: NCT07367581
Title: Costotransverse Foramen Block Versus Thoracic Paravertebral Block in Thoracotomy for Lung Cancer: A Randomized Controlled Trial
Brief Title: Costotransverse Foramen Block Versus Thoracic Paravertebral Block in Thoracotomy for Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Mai Mohamed El Rawas, Assistant professor of Anaesthesia, Intensive Care and Pain Management, National Cancer Institute, Cairo University Cairo University, Cairo, Egypt., National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP2512-501-141-205
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Costotransverse Foramen Block; Thoracic Paravertebral Block; Thoracotomy; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTFB Group (Experimental): Patients will receive an ipsilateral ultrasound-guided costotransverse foramen block with injection of 20 ml bupivacaine 0.25%.
  Interventions: Other: Costotransverse foramen block
- TPVB Group (Experimental): Patients will receive an ipsilateral ultrasound-guided thoracic paravertebral plane block with injection of 20 ml bupivacaine 0.25%.
  Interventions: Other: Thoracic paravertebral plane block

INTERVENTIONS:
Other: Costotransverse foramen block — Patients will receive an ipsilateral ultrasound-guided costotransverse foramen block with injection of 20 ml bupivacaine 0.25%.
  Arms: CTFB Group
Other: Thoracic paravertebral plane block — Patients will receive an ipsilateral ultrasound-guided thoracic paravertebral plane block with injection of 20 ml bupivacaine 0.25%.
  Arms: TPVB Group

SUMMARY:
This study aims to compare the costotransverse foramen block (CTFB) with thoracic paravertebral block (TPVB) in patients undergoing thoracotomy for lung cancer.

DETAILED DESCRIPTION:
Thoracotomy is known to be one of the most painful surgeries. Managing post-thoracotomy pain is a major clinical challenge, as about 75% of patients report moderate to severe pain afterward.

Various regional and central analgesia techniques, such as thoracic epidural analgesia (TEA), thoracic paravertebral block (TPVB), and erector spinae plane block (ESPB), are employed in a multimodal approach. Although TEA has traditionally been considered the gold standard for thoracotomy pain control, concerns about its side effects have prompted the exploration of alternatives.

The costotransverse foramen block (CTFB), a recently introduced technique, has been examined in both cadaveric and case studies.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and ≤ 65 years old.
* American Society of Anesthesiologists (ASA) physical status II-III.
* Body mass index 18-35 kg/m2.
* Patients scheduled for thoracotomies for lung cancer.

Exclusion Criteria:

* Patient refusal.
* History of sensitivity to local anesthetics.
* History of psychological disorders.
* Contraindication to regional anesthesia, e.g., local sepsis, pre-existing peripheral neuropathies, and coagulopathy.
* Severe respiratory, cardiac, hepatic, or renal disease.
* Morbid obesity.
* Uncooperative patients.
* Patients on chronic pain therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-24 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  If the visual analog scale (VAS) is ≥ 4, rescue analgesics will be administered in the form of a 4 mg bolus of morphine.

SECONDARY OUTCOMES:
Duration of analgesia | 24 hours postoperatively
  Duration of analgesia will be recorded from the end of surgery till first dose of morphine administrated.
Degree of pain | 48 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the visual analog scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). VAS will be recorded in post-anesthesia care unit (PACU) and after 1, 6, 12, 24 & 48 hours postoperatively
Intraoperative fentanyl consumption | Intraoperatively
  Intraoperative fentanyl consumption will be recorded.
Mean arterial blood pressure | 4 hours postoperatively
  Mean arterial blood pressure will be recorded before induction of general anesthesia to be defined as the baseline reading. Another reading will be noted immediately before surgical incision and at 20-minute intervals intraoperatively, and then hourly for the next 4 hours postoperatively.
Heart rate | 4 hours postoperatively
  Heart rate will be recorded before induction of general anesthesia to be defined as the baseline reading. Another reading will be noted immediately before surgical incision and at 20-minute intervals intraoperatively, and then hourly for the next 4 hours postoperatively.
Incidence of block-related side effects | 4 hours postoperatively
  Incidence of block-related side effects such as unexpected epidural anesthesia, pneumothorax, total spinal anesthesia, or local anesthetic intoxication will be recorded.
Incidence of side effects | 4 hours postoperatively
  Incidence of side effects such as postoperative nausea and vomiting, drowsiness, or dyspnea will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.